CLINICAL TRIAL: NCT06435507
Title: Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Doses of IM-250 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovative Molecules GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM-101
Record Dates: First submitted 2024-05-20; First posted 2024-05-30 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Herpes Simplex Virus
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): 6 participants
  Interventions: Drug: IM-250 (50 mg)
- Cohort 2 (Experimental): 6 participants
  Interventions: Drug: IM-250 (100 mg)
- Cohort 3 (Experimental): 6 participants
  Interventions: Drug: IM-250 (200 mg)
- Cohort 4 (Experimental): 6 participants
  Interventions: Drug: IM-250 (400 mg)

INTERVENTIONS:
Drug: IM-250 (50 mg) — Single dose
  Arms: Cohort 1
Drug: IM-250 (100 mg) — Single dose
  Arms: Cohort 2
Drug: IM-250 (200 mg) — Single dose
  Arms: Cohort 3
Drug: IM-250 (400 mg) — Single dose
  Arms: Cohort 4

SUMMARY:
This is a first-in-human, phase I, open-label, monocenter, single dose-escalation study with 4 cohorts. The total trial duration for each participant will be not more than 98 d from screening to the end of the follow-up.

Twenty-four participants are planned to be enrolled in the trial. Each cohort may be expanded by up to 6 additional volunteers, resulting in a maximum of 48 participants possibly enrolled in the trial.

Ninety-six volunteers may need to be screened to include 48 volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF),
2. Age 18-50 y inclusive at the time of consent,
3. An understanding, ability, and willingness to fully comply with study interventions and restrictions,
4. Males who are willing to use a condom for contraception during the treatment and for 60 d after IMP administration, or who are convincingly sexually abstinent, or who are refraining from heterosexual intercourse; females who are willing to use a highly effective method for contraception during the treatment and for 90 d after IMP administration, or who are convincingly sexually abstinent, or who are refraining from heterosexual intercourse, or women not of child-bearing potential (WNOCBP).
5. Satisfactory medical assessment without clinically significant or relevant abnormalities as determined by medical history, physical examination (PE), clinical (vital signs including normal heart rate [50-90 bpm]), laboratory (hematology, biochemistry, urinalysis), and electrocardiographic (ECG) evaluation (corrected QTc interval within normal range). First degree AV blocks may be acceptable, if the pulse rate complies with the inclusion criteria.
6. Ability to provide written, personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related interventions.

Exclusion Criteria:

1. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the IMP or study interventions.
2. Any intake of substances (prescription medication, over-the-counter medicine, or herbal preparations with active ingredients) known to inhibit drug-metabolizing enzymes or transport enzymes within a period of less than 5 times the respective elimination t1/2 with regard to the expected date of IMP administration (except iodine, hormone replacement therapy, hormonal contraception, and levothyroxine).
3. Any intake of substances (prescription medication, over-the-counter medicine, or herbal preparations with active ingredients) known to induce drug-metabolizing enzymes or transport enzymes within a period of 14 d with regard to the expected date of IMP administration.
4. A positive result in testing for illegal drugs at screening and enrollment.
5. Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day.
6. Consumption of alcohol within 24 h prior to Day 1 and until End of Study (EOS).
7. Clinically relevant abnormalities regarding ECG conduction (AV block), hematocrit, hemoglobin (Hb), platelets, or leucocytes. A Hb value > 12 g / dl (males) or > 11 g / dl (females) is acceptable.
8. Abnormal renal function as defined by estimated creatinine clearance: < 90 ml / min (Cockcroft-Gault equation).
9. Alanine aminotransferase (ALT) > ULN x 1.1; aspartate aminotransferase (AST) > ULN x 1.2.
10. Thyroid-stimulating hormone (TSH) not within normal limits. If thyroid hormones are supplemented, reduced TSH values are acceptable, if free thyroxine (T4) and free triiodothyronine (T3), are within the normal range.
11. Total bilirubin > upper limit of normal (ULN) x 1.2; In case of suspected Gilbert´s disease: total bilirubin ≤ ULN x 3 is acceptable.
12. Any history of severe allergic or anaphylactic reactions to drugs or food or any other clinically significant allergies.
13. Known allergy / hypersensitivity to additives used in the IMP.
14. Use of another IMP within 30 d prior to receiving the dose of IMP or active enrolment in another drug or vaccine clinical trial.
15. A positive human antibody screen for immunodeficiency virus (HIV), or chronic hepatitis C virus (HCV), or a positive hepatitis B antigen (HBsAg) test.
16. History of immunization within 14 d prior to expected dosing, including SARS-CoV-2 vaccinations, and / or plans to get vaccinated during the observation time
17. Pregnancy or breast feeding
18. Prior exposure in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Occurrence (number) of dose-limiting toxicities (DLT) | within 28 days after exposure
  * Serious adverse reaction (i.e., a serious adverse event (SAE) considered at least possibly related to IMP administration)
  * Severe (CTCAE grade III) non-serious adverse reactions (i.e., severe non-serious adverse event (AE) considered as, at least, possibly related to IMP administration) lasting more than 72 h

SECONDARY OUTCOMES:
PK: The area under the plasma concentration-time curve extrapolated to infinity (AUC∞) | 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Maximum plasma concentration (Cmax) | 8 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Concentration at 24 h (C24h), 5 d (C5d), and 8 d (C8d) | 24 hours, 5 days and 8 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)

OTHER OUTCOMES:
PK: Time to reach Cmax (Tmax) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Half-life (t1/2) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Apparent clearance (CL/F) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Mean disposition residence time (MDRT) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Volume of distribution (Vz/F) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses)
PK: Amount excreted into urine (Ae) | Follow-up 56 days
  Non-compartmental pharmacokinetic (PK) analysis (NCA) of IM-250 plasma concentrations (exposure with different doses).
  Further derived parameters may be calculated, if deemed necessary.
Safety: Description of all AE and treatment-emerging AE | Follow-up 56 days
  * System organ class (SOCs),
  * Seriousness,
  * Relatedness,
  * Severity,
  * Outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Department of Clinical Pharmacology and Pharmacoepidemiology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No